CLINICAL TRIAL: NCT00845975
Title: A Double-blind, Placebo-controlled Randomized Evaluation of the Application of Low Level Laser Light Therapy Using the Erchonia Hearing Lasers for the Relief of Tinnitus Clinical Study Protocol.
Brief Title: Study of Low Level Laser Therapy and Tinnitus Relief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New information suggested a more effective treatment protocol.
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS-001
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erchonia Hearing Lasers #1 & #2 (Active Comparator): Erchonia Hearing Laser #1 is a dual laser system composed of a pulsed red 7.5 milliwatts (mW) laser of 635 nm +/- 5 nm and a pulsed green 7.5 mW laser of 532 nm, both lasers in simultaneous operation when the laser is activated.
  Erchonia Hearing Laser #2 is a single diode laser that in pulsed mode emits 4.9 mW of red 635 nm +/- 5 nm light.
  Interventions: Device: Erchonia Hearing Lasers #1 & #2
- Placebo Lasers (Placebo Comparator): Inactive lasers that do not emit any therapeutic light.
  Interventions: Device: Placebo Lasers

INTERVENTIONS:
Device: Erchonia Hearing Lasers #1 & #2 — Two treatments with Erchonia Hearing Laser #1 administered by the investigator at the test site, each treatment seven days apart.
  Seven treatments with the Erchonia Hearing Laser #2 administered by the subject at home, one time each day for seven consecutive days, the first administration on the same day as the first administration with the Erchonia Hearing Laser #1 at the test site.
  Arms: Erchonia Hearing Lasers #1 & #2
Device: Placebo Lasers — The same test site and at-home treatment administration protocols are followed, but the laser devices do not emit any therapeutic light.
  Arms: Placebo Lasers

SUMMARY:
The purpose of this study is to determine if low level laser light therapy might help to relieve tinnitus in adults.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound, such as a ringing or hissing, that occurs in the ears or head in the absence of external stimuli. About 40-50 million people in the United States report experiencing tinnitus; 10-12 million have sought medical help for their tinnitus, with 2.5 million reporting their tinnitus as debilitating. As a result of the distressing nature of tinnitus, it is often accompanied by anxiety, depression and sleep difficulties.

Tinnitus is most often caused by sensorineural hearing loss due to presbyacusis (aging) or noise damage. It is believed that the tinnitus results when spurious neuro-electrical signals are produced by diseased, degenerated or damaged cochlear hair cells and interpreted by the brain as tinnitus.

There is presently no cure for tinnitus. Current management strategies include using other external sounds to distract from the tinnitus, teaching relaxation and stress reduction techniques, and prescription medications to help ease stress, anxiety, depression and sleep difficulties. However, in general, current tinnitus management techniques are only minimally effective. It is believed that low level laser light therapy may offer a simple, non-invasive means of relieving the symptoms of tinnitus. In theory, low level laser light penetrates targeted tissues to stimulate the mitochondria in underlying cells to produce energy through the production of adenosine triphosphate (ATP). In turn, the enhanced ATP fuels cellular energy and enhances blood flow to the cochlear hair cells (cilia) to assists in regulating the electrical signals disrupted by the diseased and/or degenerated cochlear hair cells. With the taming of the spurious electrical signals, the brain no longer has a basis to perceive the noise known as tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Total score on the Tinnitus Handicap Inventory (THI) of at least 20.
* Tinnitus is on-going; present for more than 50% of the time over the past 6 months.
* Subject has been previously evaluated by a qualified health care professional for tinnitus and received a diagnosis of etiology of tinnitus related to hearing impairment and/or noise exposure and/or unknown.
* Any existing hearing loss stable over the past 12 months.
* Willingness to abstain from partaking in other, non-study procedures indicated to lessen tinnitus and/or its perception, with the exclusion of wearing hearing aids for those subjects who enter the study using hearing aids, throughout the course of study participation.
* Willing and able to refrain from engaging in activities or work involving loud noise exposure, such as hunting, rock concerts and work situations that involve working around loud machinery, construction sites, etc., throughout the course of study participation.
* 18 years or older.
* Male or female.
* English as primary spoken language.

Exclusion Criteria:

* Presence of any of the following or in the subject's medical history:
* physical trauma or surgery to the head or neck
* uncontrolled hypertension
* current or prior surgically removed acoustic neuroma middle ear infection/active drainage from the ear and/or history of either within the previous 90 days
* impacted cerumen
* thyroid disease
* vascular disorders
* Temporomandibular Joint Disorder (TMJD)
* nutritional deficiency
* aneurysm
* multiple sclerosis
* Episodic or infrequent tinnitus
* Somatic or pulsatile tinnitus
* Prior history of sudden hearing loss and/or fluctuating hearing levels .
* Consistent use of any of the following drugs within the past 30 days:

NSAIDS; aspirin and other salicylates; Lasix and ther "loop"diuretics; "mycin" antibiotics such as vancomycin; quinine and related drugs; Chemotherapy agents such as cis-platin.

* Acute or chronic vertigo/dizziness.
* Prior diagnosis of central auditory processing disorder.
* Ménière's disease.
* Tympanic membrane perforation or tubes.
* Prior stapedectomy
* Prior mastoidectomy.
* Otosclerosis.
* Otosyphilis.
* Labyrinthitis.
* Auditory nerve damage.
* Stapedius myoclonus syndrome.
* Brain and/or brainstem injury.
* Cochlear implant.
* Photosensitivity disorder.
* Active/open infection, wound or other external trauma to the areas to be treated with the Hearing Laser.
* Pregnant or lactating.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that would make it difficult for the subject to partake in the clinical study, including adequate comprehension of the informed consent form and ability to record the necessary measurements.
* History of drug or alcohol abuse.
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to tinnitus and/or hearing loss.
* Participation in research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis A Looper, MA, CCC-A, Principal Investigator — McDonald Hearing Aid Centers
Locations (1):
- McDonald Hearing Aid Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 subjects were recruited and enrolled in this study between August 26, 2008 and September 16, 2008 at a single medical hearing aid clinic.
Pre-assignment Details: There were no significant events or approaches for the overall study following participant enrollment, but prior to group assignment. There were no enrolled participants excluded from the trial before assignment to groups.
Groups:
- Erchonia Hearing Lasers #1 & #2: Erchonia Hearing Laser #1 is a dual laser system composed of a pulsed red 7.5 milliwatts (mW) laser of 635 nm +/- 5 nm and a pulsed green 7.5 mW laser of 532 nm, both lasers in simultaneous operation when the laser is activated.
  Erchonia Hearing Laser #2 is a single diode laser that in pulsed mode emits 4.9 mW of red 635 nm +/- 5 nm light.
  Erchonia Hearing Lasers #1 & #2 : Two treatments with Erchonia Hearing Laser #1 administered by the investigator at the test site, each treatment seven days apart.
  Seven treatments with the Erchonia Hearing Laser #2 administered by the subject at home, one time each day for seven consecutive days, the first administration on the same day as the first administration with the Erchonia Hearing Laser #1 at the test site.
- Placebo Lasers: Inactive lasers that do not emit any therapeutic light.
  Placebo Lasers : The same test site and at-home treatment administration protocols are followed, but the laser devices do not emit any therapeutic light.
Period: Overall Study
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erchonia Hearing Lasers #1 & #2: Erchonia Hearing Laser #1 is a dual laser system composed of a pulsed red 7.5 mW laser of 635 nm +/- 5 nm and a pulsed green 7.5 mW laser of 532 nm, both lasers in simultaneous operation when the laser is activated.
  Erchonia Hearing Laser #2 is a single diode laser that in pulsed mode emits 4.9 mW of red 635 nm +/- 5 nm light.
  Erchonia Hearing Lasers #1 & #2 : Two treatments with Erchonia Hearing Laser #1 administered by the investigator at the test site, each treatment seven days apart.
  Seven treatments with the Erchonia Hearing Laser #2 administered by the subject at home, one time each day for seven consecutive days, the first administration on the same day as the first administration with the Erchonia Hearing Laser #1 at the test site.
- Total: Total of all reporting groups
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.53) | 66.18 (9.10) | 63.58 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Total Score on the Tinnitus Handicap Inventory (THI).
Description: The Tinnitus Handicap Inventory (THI) is a 25-item questionnaire to assess how tinnitus affects an individual's life. Each question is responded to as 'yes' (4 points); 'sometimes' (2 points) or 'no' (0 points). The individual scores for the 25 questions are added to get a total THI score from 0 to 100. The higher the total THI score, the greater the negative impact tinnitus has on the individual's life. Change in total THI score is calculated as total THI score after the one week procedure administration phase minus total THI score at baseline. A positive (+) change in total THI score indicates the negative impact of tinnitus on the individual's everyday life has worsened. A negative (-) change indicates the negative impact of tinnitus on the individual's everyday life has improved (lessened). A change in total THI score of -20 or greater indicates a meaningful lessening of the impact of tinnitus on the individual's life and is positive for study success.
Time Frame: baseline and one week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers
Number analyzed (Participants) | 9 | 9
units on a scale | -22.80 (18.63) | -16.66 (13.48)

2. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The Beck Depression Inventory®-II (BDI®-II) is a 21-item questionnaire used to assess depression. Most items are rated on a 4-point scale from 0 to 3, and a few items are rated on a 7-point scale. Individual item scores are added to get a total score from 0 to 63. The higher the total score, the more severe the depression, and the lower the total score, the less severe the depression. Change in BDI®-II score is calculated as the BDI®-II score 4 weeks after baseline evaluation minus the BDI®-II score at baseline. A positive (+) change in BDI®-II score indicates that the depression has worsened. A negative (-) change in BDI®-II score indicates the depression has lessened. A change in BDI®-II score of -6 or greater indicates a meaningful lessening of depression and is positive for study success.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers
Number analyzed (Participants) | 9 | 9
units on a scale | -4.3 (3.56) | -2.5 (1.98)

3. Secondary Outcome: Spielberger State-Trait Anxiety Inventory (STAI)- Trait Portion
Description: The Trait portion of the State-Trait Anxiety Inventory (STAI-T) evaluates an individual's tendency to get anxious and how they respond to stress. The STAI-T has 20 items rated on a 4-point frequency of occurrence scale of 1=Almost Never, 2=Sometimes, 3=Moderately So, and 4=Very Much So. The individual scores are summed to get the total STAI-T score. The higher the total score, the more anxious the individual, and the lower the total score, the less anxious the individual. Change in STAI-T score is calculated as the STAI-T score at 4 weeks after baseline evaluation minus the STAI-T score at baseline. A positive (+) change in STAI-T score indicates that the anxiety has worsened. A negative (-) change in STAI-T score indicates the depression has lessened. A change in STAI-T score of -8 or greater indicates a meaningful lessening of anxiety and is positive for study success.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers
Number analyzed (Participants) | 9 | 9
units on a scale | -0.2 (1.32) | -2.88 (3.45)

ADVERSE EVENTS:
Arm/Group | Erchonia Hearing Lasers #1 & #2 | Placebo Lasers
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No